CLINICAL TRIAL: NCT02072382
Title: The Hypotensive Effect of Simvastatin in Hypertensive Patients: a Placebo-controlled Randomized Clinical Trial With 24-h Ambulatory Blood Pressure Monitoring
Brief Title: The Hypotensive Effect of Metformin in Hypertensive Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 120406
Record Dates: First submitted 2013-09-16; First posted 2014-02-26 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Hypertension
Keywords: Hypertension; Metformin; Ambulatory blood pressure monitor
MeSH Terms: conditions — Hypertension | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin (Experimental): Metformin 850 mg twice a day for eight weeks versus Placebo
  Interventions: Drug: Metformin; Drug: Placebo

INTERVENTIONS:
Drug: Metformin — metformin 850mg twice a day for eight weeks
  Other Names: Glucophage
Drug: Placebo

SUMMARY:
The proposed study is to evaluate the possible effect of metformin on arterial pressure by 24h-ambulatory blood pressure monitory (24h-ABPM).

DETAILED DESCRIPTION:
The primary outcome was the difference in mean 24-hour blood pressure variation between the two groups after the intervention. The difference in mean of blood pressure during daytime and nighttime in 24h ambulatory blood pressure monitory, as well as the office BP and laboratory differences were considered secondary outcomes.

This randomized, double-blind parallel study was conducted in the Hypertension Clinic of the Department of Cardiology, Hospital de Clínicas de Porto Alegre (Porto Alegre, Brazil).

We selected hypertensive individuals (controlled or not) without diabetes aged 18-70 years.

Exclusion criteria: metformin intolerance, creatinine > 1,5 mg/dl Risks: adverse effects related to metformin use, mainly diarrhea and nausea Benefits: possible lower effect on arterial pressure Statistical analysis: sample size was calculated on the basis of a standard deviation of 8 mm Hg and effect size of 5 mm Hg in 24-h systolic ABPM and a two-sided significance level of 5%. A sample size of 42 patients per group was estimated to provide a power of 80% to reject the null hypothesis. Considering possible 10% of losses, the final calculated sample was 92 patients.

The baseline comparison between groups was performed using the Student t test for continuous variables and x2 for categorical variables. In each group, the change in BP by ABPM -24 h, daytime and nighttime, and laboratory tests was calculated by subtracting baseline values measured after the intervention period. The difference between groups was calculated by subtracting the variation observed between them (δ-values). The differences in BP variation and laboratory tests were analyzed by analysis of variance for repeated measures (MANOVA). For differences in pressure variation adjustment was considered for the baseline BP values (analysis of covariance). All tests were two-tailed and significance level was 5%. Data were analyzed using Statistical Package for the Social Sciences (SPSS) version 13.0.

ELIGIBILITY:
Inclusion Criteria:

* hypertensive patients,
* aged 18-75 years

Exclusion Criteria:

* diabetes
* metformin intolerance
* creatinine level above 1.5 mg/dL

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The effect of metformin on blood pressure | eight weeks
  The primary outcome was the difference in mean 24-hour BP variation between the two groups (metformin versus placebo) after the intervention.

SECONDARY OUTCOMES:
The difference in mean of BP during daytime and nighttime in ABPM-24h, as well as the office BP and laboratory differences were considered secondary outcomes. | eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gus Miguel, Study Chair — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil